CLINICAL TRIAL: NCT00061308
Title: An Open-label, Multicenter, Non-Comparative Phase II Study of the Combination of Intravenous Topotecan and Gemcitabine Administered Once Weekly for Three Weeks Every 28 Days as Second-line Treatment in Patients With Recurrent Platinum Sensitive Ovarian Cancer
Brief Title: Second-line Intravenous Treatment For Recurrent Platinum-Sensitive Ovarian, Fallopian, Or Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 104864/627
Record Dates: First submitted 2003-05-23; First posted 2003-05-28 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2013-03

CONDITIONS: Peritoneal Cancer; Ovarian Cancer; Neoplasms, Ovarian; Fallopian Tube Cancer
Keywords: Ovarian cancer; peritoneal cancer; cancer; Fallopian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Neoplasms | interventions — Topotecan; Gemcitabine

INTERVENTIONS:
Drug: Topotecan
Drug: Gemcitabine
  Other Names: Topotecan

SUMMARY:
This research study was designed to determine the effectiveness of the drug, topotecan, given intravenously (into a vein) together with the drug gemcitabine in patients with recurrent platinum-sensitive ovarian, fallopian or primary peritoneal cancer, as well as tumors of mixed mullerian origin. Additional purposes are to determine the long term outcome and side effects of this combination treatment.

Since topotecan and gemcitabine have different mechanisms of action, the combination of these 2 drugs may provide better results than either drug alone. Prior studies suggest that the combination of topotecan and gemcitabine improves the effects on the tumor and also appeared to be well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Have had one prior platinum-based chemotherapy regimen for the treatment of primary disease.
* At least 4 weeks since last surgery or radiation therapy.
* Must have had a treatment-free interval of greater than 6 months following response to platinum.
* ECOG performance status of 0,1, or 2.

Exclusion Criteria:

* Women of child-bearing potential that do not practice adequate contraception.
* Pregnant or lactating.
* Received more than one primary chemotherapy regimen.
* Concomitant or previous malignancies with the exception of adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, incidental carcinoid, or other cancer from which the patient has been disease free for 5 years.
* Active uncontrolled infection requiring antibiotics.
* Concurrent severe medical problems unrelated to the malignancy which would limit full compliance with the study.
* Received radiation to more than 10% of bone.
* Prior treatment with topotecan or gemcitabine.
* Hypersensitivity to camptothecin or nucleoside analogues.
* Use of an investigational agent within 30 days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2002-12; Primary Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
response rate

SECONDARY OUTCOMES:
response duration time to response time to progression survival safety

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, PhD, Study Director — GlaxoSmithKline
Locations (19):
- United States (15):
  - GSK Investigational Site, Los Gatos, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Hinsdale, Illinois
  - GSK Investigational Site, Lansing, Michigan
  - GSK Investigational Site, Southfield, Michigan
  - GSK Investigational Site, Hattiesburg, Mississippi
  - GSK Investigational Site, Saint Louis, Montana
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Abington, Pennsylvania
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario

REFERENCES:
- See also: A website where viewers can complete a clinical study-matching questionnaire and also sign up for future study notification and healthcare newsletters. — http://www.findclinicalstudy.com